CLINICAL TRIAL: NCT00415142
Title: An Eight-week, Multinational, Multicenter, Randomized, Double-blind, Placebo-controlled Study, With Escitalopram as an Active Control, to Evaluate the Efficacy, Safety and Tolerability of a Saredutant 100 mg Dose Once Daily, in Elderly Patients With Major Depressive Disorder
Brief Title: An Eight-week Study Evaluating the Efficacy of a 100mg Dose of Saredutant Once Daily, in Elderly Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5574
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Depressive Disorder
Keywords: Depression; Major depressive disorders; Controlled clinical trial
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major | interventions — SR 48968; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saredutant 100 mg (Experimental): Saredudant100 mg once daily for a maximum of 32 weeks
  Interventions: Drug: saredutant (SR48968)
- Escitalopram 10 mg (Active Comparator): Escitalopram 10 mg once daily for a maximum of 32 weeks
  Interventions: Drug: escitalopram
- Placebo (Placebo Comparator): Placebo once daily for one week during screening phase and a maximum of 8 weeks during the acute phase
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: saredutant (SR48968) — oral administration (capsules)
  Arms: Saredutant 100 mg
Drug: placebo — oral administration (capsules)
  Arms: Placebo
Drug: escitalopram — oral administration (capsules)
  Arms: Escitalopram 10 mg

SUMMARY:
The purpose of the study is to evaluate the efficacy of saredutant in the treatment of Major Depressive Disorder in elderly patients.To evaluate the tolerability, safety and efficacy on disability and quality of life in patients with major depressive disorder.To evaluate safety and tolerability of 24 weeks of additional treatment in patients completing the initial 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder, recurrent, as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) criteria (296.3) and confirmed by the semi-structured Mini International Neuropsychiatric Interview (MINI).

Exclusion Criteria:

* Total score of less than 23 on the MADRS.
* HAM-D total score less than 17.
* Duration of the current depressive episode less than 1 month or greater than 2 years.
* Patients with an Mini Mental State Examination score of less than 23.
* Patients with a history or presence of bipolar disorders or psychotic disorders.
* Patients with alcohol/substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* Patients who have used the following prior to entry into Acute Phase: antipsychotics within 3 months, fluoxetine within 1 month, monoamine oxidase inhibitors within 4 weeks, other antidepressants, or mood-stabilizer (lithium, anticonvulsants) within 1 week.

The investigator will evaluate whether there are other reasons why a patient may not participate

Ages: 60 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 393 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 56 in the 17-item Hamilton Depression Rating Scale (HAM-D) total score. | Day 56

SECONDARY OUTCOMES:
Change from baseline to Day 56 in the Clinical Global Impression (CGI) Severity of Illness score. | Day 56
Change from baseline to Day 56 in the HAM-D depressed mood item score | Day 56
Change from baseline to Day 56 in the Montgomery-Asberg Depression Rating Scale (MADRS) total score | Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)